CLINICAL TRIAL: NCT02010229
Title: Clinical Situations at High Risk of Placenta Accreta / Percreta: Impact of Diagnostic Methods and Management on Maternal Morbidity.
Brief Title: Clinical Situations at High Risk of Placenta Accreta / Percreta
Acronym: Paccreta
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Inserm U953 (Epidemiological research unit on perinatal health and women's and children's health) Paris, France (Unknown); University Hospital, Angers (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI11061
Record Dates: First submitted 2013-11-21; First posted 2013-12-12 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Placenta Accreta / Percreta
Keywords: Placenta accreta; previous caesarean; placenta praevia; severe obstetric haemorrhage; population-based study
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women at high risk of placenta accreta: Parturient women with placenta praevia and at least one previous caesarean delivery

SUMMARY:
The purpose of this study is to identify what factors -either individual or related to the type of management received- influence the maternal outcomes in pregnant women at high risk for placenta accreta i.e , women with placenta praevia and previous caesarean.

This population-based study conducted in 8 French regions will also provide valid estimation of the incidence of placenta accreta among all parturients and among "at risk "women. Finally, a psychological evaluation of these women up to 1 year after delivery will provide information on the impact of these conditions on women, beyond somatic complications.

DETAILED DESCRIPTION:
Background: No population-based study has assessed the prevalence of placenta accreta, the predictive value of prenatal diagnostic examinations, the maternal morbidity associated with its management, or its psychological effects. Moreover the technical resources necessary for the safest delivery of women at risk have not been clearly identified.

Objectives: The primary objectives are to identify individual risk factors for maternal morbidity, as well as risk factors related to types of management and healthcare facilities for postpartum hemorrhage (PPH). Secondary objectives are to 1) determine the prevalence of placenta accreta among women at risk; 2) assess the predictive value of ultrasound and MRI for the diagnosis of placenta accreta in this population; 3) evaluate psychological impact and physical complications; 4) report maternal physical complications during the year after delivery.

Design: Population-based prospective observational study of pregnant women with a placenta inserted at a uterine scar Setting; A total of 166 centers in 8 French regions, with 260,000 deliveries annually.

Methods: We expect to include 570 women at risk of placenta accreta in two years, of whom approximately 100 (20%) will have placenta accreta.

Main outcome measures: The primary outcome measure is severe maternal hemorrhage; secondary outcome measures are maternal morbidity and deaths, predictive value of ultrasound and MRI, and psychological evaluations at 1, 6 and 12 months after delivery.

Conclusion: This study will be the first prospective population-based study to include women at risk of placenta accreta and to investigate incidence, prenatal detection, type of management, morbidity and maternal psychological consequences.

ELIGIBILITY:
Inclusion Criteria:

Every woman:

* delivering in a maternity unit of the 11 participating perinatal networks.
* With a placenta praevia and at least one previous cesarean delivery, and / or having a placenta accreta
* aged 18 or more

Exclusion Criteria:

Every woman:

* not understanding French.
* refusing to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women delivering in maternity units of 8 French regions.
Sampling Method: Non-Probability Sample
Enrollment: 674 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Severe postpartum hemorrhage | up to 7 days post delivery
  Severe hemorrhage defined by a hemorrhage with transfusion of at least four red blood cell units.

SECONDARY OUTCOMES:
Incidence of accreta or percreta placenta overall and in women with previous caesarean section and placenta praevia | At delivery
  Number of women with placenta accreta divided 1)by the number of parturient women, and 2) by the number of women with previous caesarean section and placenta praevia
Predictive value of prenatal ultrasound and MRI for the diagnosis of placenta accreta in women with previous caesarean section and placenta praevia | at delivery
  Sensitivity, specificity and positive and negative predictive values.
severe maternal morbidity | up to 6 months post-delivery
  haemorrhage, infection, intraoperative and postoperative complications, thromboembolic complications.
Psychological impact | at 1 year post-delivery
  All the women will receive several validated auto-questionnaires (postpartum depression, anxiety, post-traumatic stress).
Psychological impact | at 1 month post-delivery
  All the women will receive several validated auto-questionnaires (postpartum depression, anxiety, post-traumatic stress)
Psychological impact | at 6 month post-delivery
  All the women will receive several validated auto-questionnaires (postpartum depression, anxiety, post-traumatic stress)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Kayem, MD, PhD, Principal Investigator — Louis Mourier University Hospital (APHP), department of gynaecology and obstetrics, Colombes, France; Loic Sentilhes, MD, PhD, Principal Investigator — Angers University Hospital, department of gynaecology and obstetrics, France; Catherine Deneux-Tharaux, MD, PhD, Study Director — INSERM U953, Epidemiological research unit on perinatal health and children's and women's health, Paris, France
Locations (1):
- Hôpital Louis Mourier (APHP), Colombes, France

REFERENCES:
- [Result] Sentilhes L, Seco A, Azria E, Beucher G, Bonnet MP, Branger B, Carbillon L, Chiesa C, Crenn-Hebert C, Dreyfus M, Dupont C, Fresson J, Huissoud C, Langer B, Morel O, Patrier S, Perrotin F, Raynal P, Rozenberg P, Rudigoz RC, Vendittelli F, Winer N, Deneux-Tharaux C, Kayem G; PACCRETA Study Group. Conservative management or cesarean hysterectomy for placenta accreta spectrum: the PACCRETA prospective study. Am J Obstet Gynecol. 2022 Jun;226(6):839.e1-839.e24. doi: 10.1016/j.ajog.2021.12.013. Epub 2021 Dec 14. PMID 34914894